CLINICAL TRIAL: NCT03858673
Title: Comparison of the Vault Prolapse Rate After Vaginal Hysterectomy With or Without Residual Uterine Ligament Ligation
Brief Title: Comparison of PHVP of Different VTH Methods
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201601062RINA
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2016-02

CONDITIONS: Vault Prolapse, Vaginal
Keywords: Vault prolapse; Vaginal total hysterectomy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ligations group: VTH via the Tsuzi method with residual uterine ligament ligation (ligations group)
  Interventions: Procedure: VTH via the Tsuzi method with residual uterine ligament ligation
- Without ligations group: Traditional VTH without residual uterine ligament ligation (without ligations group)

INTERVENTIONS:
Procedure: VTH via the Tsuzi method with residual uterine ligament ligation — VTH via the Tsuzi method with residual uterine ligament ligation
  Groups: Ligations group

SUMMARY:
To evaluate the post-hysterectomy vault prolapse (PHVP) rates performed using different methods of vaginal total hysterectomy (VTH).

DETAILED DESCRIPTION:
Objective: To evaluate the post-hysterectomy vault prolapse (PHVP) rates performed using different methods of vaginal total hysterectomy (VTH).

Methods: A computer search identified a total of 251 women who underwent VTH with/without concomitant surgeries between January 1986 and December 2001 in a single center. Thirty-eight women were excluded due to not only a vaginal approach. Of the remaining 213 women, 129 and 84 underwent VTH via the Tsuzi method with residual uterine ligament ligation (ligations group) and traditional VTH (without ligations group), respectively. The χ2 and Mann-Whitney U tests were applied to compare the data. The cumulative percentages of women without PHVP were calculated over time and compared using Kaplan-Meier curves and log-rank tests. A p value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Received VTH with or without other combined operations.

Exclusion Criteria:

1. Laparoscopic-assisted vaginal hysterectomy (LAVH)
2. Conversion to an abdominal approach
3. Unsatisfactory medical record

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 1986 and December 2001, all women who received VTH with or without other combined operations at National Taiwan University Hospital were recruited. In September 2016, a retrospective chart review was performed.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 1986-01-01 (Actual); Primary Completion 2001-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Post-hysterectomy vault prolapse | Between January 1986 and December 2001
  PHVP was defined as more than or equal to the second stage of descent of the vaginal vault was noted during the follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Result] Buca DIP, Liberati M, Falo E, Leombroni M, Di Giminiani M, Di Nicola M, Santarelli A, Frondaroli F, Fanfani F. Long-term outcome after surgical repair of pelvic organ prolapse with Elevate Prolapse Repair System. J Obstet Gynaecol. 2018 Aug;38(6):854-859. doi: 10.1080/01443615.2017.1419462. Epub 2018 Mar 14. PMID 29537324
- [Result] Ker CR, Lin KL, Loo ZX, Juan YS, Long CY. Comparison of UpholdTM Vaginal Mesh Procedure with Hysterectomy or Uterine Preservation for the Treatment of Pelvic Organ Prolapse. Sci Rep. 2018 Jun 21;8(1):9438. doi: 10.1038/s41598-018-27765-8. PMID 29930249
- [Result] Chang TC, Hsiao SM, Chen CH, Wu WY, Lin HH. Clinical Outcomes and Urodynamic Effects of Tailored Transvaginal Mesh Surgery for Pelvic Organ Prolapse. Biomed Res Int. 2015;2015:191258. doi: 10.1155/2015/191258. Epub 2015 Nov 8. PMID 26634203
- [Result] Chen CH, Hsiao SM, Chang TC, Wu WY, Lin HH. Transvaginal cystocele repair using pursestring technique reinforced with custom-tailored two-armed mesh. Urology. 2011 Dec;78(6):1275-80. doi: 10.1016/j.urology.2011.07.1380. Epub 2011 Sep 9. PMID 21908027